CLINICAL TRIAL: NCT03942328
Title: MC1641 Phase II Study Of Intratumoral Injection Of Autologous Dendritic Cells Combined With Immune Checkpoint Inhibition After High-Dose Conformal External Beam Radiotherapy In Patients With Unresectable Primary Liver Cancer
Brief Title: Modified Immune Cells (Autologous Dendritic Cells) and a Vaccine (Prevnar) Combined With Immune Checkpoint Inhibition After High-Dose External Beam Radiation Therapy in Treating Patients With Unresectable Liver Cancer
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: MC1641; R01CA274985 (NIH); R01CA294704 (NIH); NCI-2019-02452 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 16-009335 (Other: Mayo Clinic Institutional Review Board)
Record Dates: First submitted 2019-05-06; First posted 2019-05-08 (Actual); Last update posted 2025-09-29 (Actual); Status verified 2025-09

CONDITIONS: Stage III Hepatocellular Carcinoma AJCC v8; Stage III Intrahepatic Cholangiocarcinoma AJCC v8; Stage IV Hepatocellular Carcinoma AJCC v8; Stage IV Intrahepatic Cholangiocarcinoma AJCC v8; Unresectable Hepatocellular Carcinoma; Unresectable Intrahepatic Cholangiocarcinoma
MeSH Terms: conditions — Carcinoma, Hepatocellular; Cholangiocarcinoma | interventions — atezolizumab; Bevacizumab; Immunoglobulin G; Disulfides; Congresses as Topic; Radiation; Blood Component Removal; 13-valent pneumococcal vaccine; Tiragolumab; Endoscopy, Digestive System; Gastroscopy; Magnetic Resonance Spectroscopy; Biopsy; Specimen Handling

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Phase II Group 2 (EBRT, dendritic cells, Prevnar, atezo, bev) (Experimental): Patients with unresectable HCC undergo apheresis for dendric cell manufacturing and standard of care high-dose EBRT for 5 or 15 fractions over 1-3 weeks (cycle 1). Patients then receive autologous dendritic cells IT on day 1 of cycles 2-8 and pneumococcal 13-valent conjugate vaccine or other pneumococcal vaccine IM on day 1 of cycles 2-4 only. Patients also receive standard of care atezolizumab IV over 30-60 minutes and bevacizumab IV over 30-90 minutes starting on day 2 of cycles 2-8. Treatment repeats every 21 days for up to 7 cycles in the absence of disease progression or unacceptable toxicity. Additionally, patients undergo an EGD at screening and CT, PET/CT and/or MRI, biopsy and urine and blood sample collection throughout the study.
  Interventions: Biological: Atezolizumab; Biological: Bevacizumab; Radiation: External Beam Radiation Therapy; Procedure: Pheresis; Biological: Pneumococcal 13-valent Conjugate Vaccine; Biological: Therapeutic Autologous Dendritic Cells; Procedure: Esophagogastroduodenoscopy; Procedure: Computed Tomography; Procedure: Positron Emission Tomography; Procedure: Magnetic Resonance Imaging; Procedure: Biopsy Procedure; Procedure: Biospecimen Collection
- Pilot study (pheresis, EBRT, dendritic cells, Prevnar) (Experimental): Patients with unresectable intrahepatic CCA undergo apheresis for dendric cell manufacturing and standard of care high-dose EBRT for 5 or 15 fractions over 1-3 weeks (cycle 1). Patients then receive autologous dendritic cells IT on day 1 of cycles 2-8 and pneumococcal 13-valent conjugate vaccine IM on day 1 of cycles 2-4 only. Treatment repeats every 28 days for up to 7 cycles in the absence of disease progression or unacceptable toxicity. (CLOSED WITH AMENDMENT 3)
  Interventions: Radiation: External Beam Radiation Therapy; Procedure: Pheresis; Biological: Pneumococcal 13-valent Conjugate Vaccine; Biological: Therapeutic Autologous Dendritic Cells
- Phase II Group 3 (EBRT, dendritic cells, Prevnar, atezo, tir) (Experimental): Patients with iCCA undergo apheresis for dendric cell manufacturing and standard of care high-dose EBRT for 5 or 15 fractions over 1-3 weeks (cycle 1). Patients then receive autologous dendritic cells IT on day 1 of cycles 2-8 and pneumococcal 13-valent conjugate vaccine or other pneumococcal vaccine IM on day 1 of cycles 2-4 only. Patients also receive standard of care atezolizumab IV over 30-60 minutes and tiragolumab IV over 30-60 minutes starting on day 2 of cycles 2-8. Treatment repeats every 21 days for up to 7 cycles in the absence of disease progression or unacceptable toxicity. Additionally, patients undergo CT, PET/CT and/or MRI, biopsy and urine and blood sample collection throughout the study.
  Interventions: Biological: Atezolizumab; Radiation: External Beam Radiation Therapy; Procedure: Pheresis; Biological: Pneumococcal 13-valent Conjugate Vaccine; Biological: Therapeutic Autologous Dendritic Cells; Biological: Tiragolumab; Procedure: Computed Tomography; Procedure: Positron Emission Tomography; Procedure: Magnetic Resonance Imaging; Procedure: Biopsy Procedure; Procedure: Biospecimen Collection

INTERVENTIONS:
Biological: Atezolizumab — Given IV
  Other Names: MPDL 3280A; MPDL 328OA; MPDL-3280A; MPDL3280A; MPDL328OA; RG7446; RO5541267; Tecentriq
  Arms: Phase II Group 2 (EBRT, dendritic cells, Prevnar, atezo, bev); Phase II Group 3 (EBRT, dendritic cells, Prevnar, atezo, tir)
Biological: Bevacizumab — Given IV
  Other Names: ABP 215; Anti-VEGF; Anti-VEGF Humanized Monoclonal Antibody; Anti-VEGF Monoclonal Antibody SIBP04; Anti-VEGF rhuMAb; Avastin; Bevacizumab awwb; Bevacizumab Biosimilar ABP 215; Bevacizumab Biosimilar BEVZ92; Bevacizumab Biosimilar BI 695502; Bevacizumab Biosimilar CBT 124; Bevacizumab Biosimilar CT-P16; Bevacizumab Biosimilar FKB238; Bevacizumab Biosimilar GB-222; Bevacizumab Biosimilar HD204; Bevacizumab Biosimilar HLX04; Bevacizumab Biosimilar IBI305; Bevacizumab Biosimilar LY01008; Bevacizumab Biosimilar MIL60; Bevacizumab Biosimilar Mvasi; Bevacizumab Biosimilar MYL-1402O; Bevacizumab Biosimilar QL 1101; Bevacizumab Biosimilar QL1101; Bevacizumab Biosimilar RPH-001; Bevacizumab Biosimilar SCT501; Bevacizumab Biosimilar Zirabev; Bevacizumab-awwb; Bevacizumab-bvzr; BP102; BP102 Biosimilar; HD204; Immunoglobulin G1 (Human-Mouse Monoclonal rhuMab-VEGF Gamma-Chain Anti-Human Vascular Endothelial Growth Factor), Disulfide With Human-Mouse Monoclonal rhuMab-VEGF Light Chain, Dimer; Mvasi; MYL-1402O; QL1101; Recombinant Humanized Anti-VEGF Monoclonal Antibody; rhuMab-VEGF; SCT501; SIBP 04; SIBP-04; SIBP04; Zirabev; Alymsys; Avzivi; Aybintio; Onbevzi; Oyavas; Vegzelma
  Arms: Phase II Group 2 (EBRT, dendritic cells, Prevnar, atezo, bev)
Radiation: External Beam Radiation Therapy — Undergo high-dose EBRT
  Other Names: Definitive Radiation Therapy; EBRT; External Beam Radiation; External Beam Radiotherapy; External Beam Radiotherapy (conventional); External Beam RT; external radiation; External Radiation Therapy; external-beam radiation; Radiation, External Beam; Teleradiotherapy; Teletherapy; Teletherapy Radiation
Procedure: Pheresis — Undergo apheresis
  Other Names: Apheresed; Apheresis; Blood Component Removal; Collection, Apheresis/Leukapheresis; Hemapheresis
Biological: Pneumococcal 13-valent Conjugate Vaccine — Given IM
  Other Names: PCV 13; PCV13 Vaccine; Prevnar 13
Biological: Therapeutic Autologous Dendritic Cells — Given IT
Biological: Tiragolumab — Given IV
  Other Names: 1918185-84-8; MTIG7192A; RG6058
  Arms: Phase II Group 3 (EBRT, dendritic cells, Prevnar, atezo, tir)
Procedure: Esophagogastroduodenoscopy — Undergo EGD
  Other Names: EGD; Upper Endoscopy
  Arms: Phase II Group 2 (EBRT, dendritic cells, Prevnar, atezo, bev)
Procedure: Computed Tomography — Undergo CT or PET/CT
  Other Names: CAT; CAT Scan; Computed Axial Tomography; computerized axial tomography; computerized tomography; Computerized Tomography (CT) scan; CT; CT SCAN; Diagnostic CAT Scan
  Arms: Phase II Group 2 (EBRT, dendritic cells, Prevnar, atezo, bev); Phase II Group 3 (EBRT, dendritic cells, Prevnar, atezo, tir)
Procedure: Positron Emission Tomography — Undergo PET/CT
  Other Names: Medical Imaging, Positron Emission Tomography; PET; PET Scan; positron emission tomography scan; PT
  Arms: Phase II Group 2 (EBRT, dendritic cells, Prevnar, atezo, bev); Phase II Group 3 (EBRT, dendritic cells, Prevnar, atezo, tir)
Procedure: Magnetic Resonance Imaging — Undergo MRI
  Other Names: MRI; Magnetic Resonance Imaging (MRI); Medical Imaging, Magnetic Resonance / Nuclear Magnetic Resonance; MR; NMRI; Nuclear Magnetic Resonance Imaging; sMRI; Structural MRI
  Arms: Phase II Group 2 (EBRT, dendritic cells, Prevnar, atezo, bev); Phase II Group 3 (EBRT, dendritic cells, Prevnar, atezo, tir)
Procedure: Biopsy Procedure — Undergo biopsy
  Other Names: BIOPSY; Bx
  Arms: Phase II Group 2 (EBRT, dendritic cells, Prevnar, atezo, bev); Phase II Group 3 (EBRT, dendritic cells, Prevnar, atezo, tir)
Procedure: Biospecimen Collection — Undergo urine and blood sample collection
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
  Arms: Phase II Group 2 (EBRT, dendritic cells, Prevnar, atezo, bev); Phase II Group 3 (EBRT, dendritic cells, Prevnar, atezo, tir)

SUMMARY:
This early phase I trial studies the side effects of autologous dendritic cells and a vaccine called Prevnar in combination with immune checkpoint inhibition (with bevacizumab and atezolizumab or atezolizumab and tiragolumab) in treating patients liver cancer that cannot be removed by surgery (unresectable) after undergoing standard high-dose external beam radiotherapy. Autologous dendritic cells are immune cells generated from patients' own white blood cells that are grown in a special lab and trained to stimulate the immune system to destroy tumor cells. A pneumonia vaccine called Prevnar may also help stimulate the immune system. Bevacizumab is in a class of medications called antiangiogenic agents. It works by stopping the formation of blood vessels that bring oxygen and nutrients to tumor. This may slow the growth and spread of tumor. Immunotherapy with monoclonal antibodies, such as atezolizumab and tiragolumab, may help the body's immune system attack the tumor, and may interfere with the ability of tumor cells to grow and spread. Giving autologous dendritic cells and Prevnar in combination with immune checkpoint inhibition after radiotherapy may be safe, and tolerable and may stimulate the body's own immune system to fight against the tumor in patients with unresectable liver cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. Evaluation of safety and tolerability of an autologous dendritic cell (DC) vaccine delivered by intra-tumoral injection in patients with primary liver cancer treated with high-dose conformal external beam radiotherapy (EBRT). (Pilot Study) II. Estimate the progression-free survival rate at 2 years post-registration to see if treatment is efficacious compared to historical data in hepatocellular carcinoma (HCC). (Phase II Group 2) II. Estimate the progression-free survival to see if treatment is efficacious compared to historical data in intrahepatic cholangiocarcinoma (iCCA) patients. (Phase II Group 3)

SECONDARY OBJECTIVES:

I. To assess feasibility in patients with liver cancer treated with high-dose conformal EBRT followed by autologous DC vaccine injection by group (Group 1 versus [vs.] 2 vs. 3).

II. To assess overall response rate in patients with liver cancer treated with high-dose conformal EBRT followed by autologous DC vaccine injection by group (Group 1 vs. 2 vs. 3).

III. To assess progression free survival in patients with liver cancer treated with high-dose conformal EBRT followed by autologous DC vaccine injection by group (Group 1 vs. 2 vs. 3).

IV. To assess clinical benefit rate in patients with liver cancer treated with high-dose conformal EBRT followed by autologous DC vaccine injection by group (Group 1 vs. 2 vs. 3).

V. To assess time to response in patients with liver cancer treated with high-dose conformal EBRT followed by autologous DC vaccine injection by group (Group 1 vs. 2 vs. 3).

VI. To assess duration of response in patients with liver cancer treated with high-dose conformal EBRT followed by autologous DC vaccine injection by group (Group 1 vs. 2 vs. 3).

VII. To assess overall survival in patients with liver cancer treated with high-dose conformal EBRT followed by autologous DC vaccine injection by group (Group 1 vs. 2 vs. 3).

RADIOLOGIC STUDY OBJECTIVE:

I. To assess the radiologic response over time of primary liver tumors treated with high-dose conformal EBRT followed by autologous DC vaccine injection by group (Group 1 vs. 2 vs. 3).

CORRELATIVE RESEARCH OBJECTIVES:

I. To monitor patients' immune response after vaccine therapy by group (Group 1 vs. 2 vs. 3).

II. To assess the immune response to pneumococcal 13-valent conjugate vaccine (Prevnar) and similar pneumococcal vaccines by group (Group 1 vs. 2 vs. 3).

OUTLINE:

PILOT STUDY (GROUP I) (CLOSED WITH AMENDMENT 3): Patients with unresectable intrahepatic cholangiocarcinoma (CCA) undergo apheresis for dendric cell manufacturing and standard of care high-dose EBRT for 5 or 15 fractions over 1-3 weeks (cycle 1). Patients then receive autologous dendritic cells intratumorally (IT) on day 1 of cycles 2-8 and pneumococcal 13-valent conjugate vaccine intramuscularly (IM) on day 1 of cycles 2-4 only. Treatment repeats every 28 days for up to 7 cycles in the absence of disease progression or unacceptable toxicity.

PHASE II STUDY (GROUP II): Patients with unresectable HCC undergo apheresis for dendric cell manufacturing and standard of care high-dose EBRT for 5 or 15 fractions over 1-3 weeks (cycle 1). Patients then receive autologous dendritic cells IT on day 1 of cycles 2-8 and pneumococcal 13-valent conjugate vaccine or other pneumococcal vaccine IM on day 1 of cycles 2-4 only. Patients also receive standard of care atezolizumab intravenously (IV) over 30-60 minutes and bevacizumab IV over 30-90 minutes starting on day 2 of cycles 2-8. Treatment repeats every 21 days for up to 7 cycles in the absence of disease progression or unacceptable toxicity. Additionally, patients undergo an esophagogastroduodenoscopy (EGD) at screening and CT, PET/CT and/or MRI, biopsy and urine and blood sample collection throughout the study.

PHASE II STUDY (GROUP III): Patients with iCCA undergo apheresis for dendric cell manufacturing and standard of care high-dose EBRT for 5 or 15 fractions over 1-3 weeks (cycle 1). Patients then receive autologous dendritic cells IT on day 1 of cycles 2-8 and pneumococcal 13-valent conjugate vaccine or other pneumococcal vaccine IM on day 1 of cycles 2-4 only. Patients also receive standard of care atezolizumab IV over 30-60 minutes and tiragolumab IV over 30-60 minutes starting on day 2 of cycles 2-8. Treatment repeats every 21 days for up to 7 cycles in the absence of disease progression or unacceptable toxicity. Additionally, patients undergo CT, PET/CT and/or MRI, biopsy and urine and blood sample collection throughout the study.

After completion of study treatment, patients are followed up at 2 weeks and then every 3 months for 1 year (beginning at week 36 or 12 weeks after last autologous dendritic cell dose whichever is earlier). Patients are then followed every 3 months until disease progression, and then every 6 months until 5 years after registration.

ELIGIBILITY:
Inclusion Criteria:

* Age >= 18 years
* Pilot study (group 1): Histologic confirmation of intrahepatic CCA (Closed as of amendment 3)
* Phase II study (group 2): Histologic and/or radiologic confirmation of hepatocellular carcinoma (HCC)
* Phase II study (group 3): Histologic confirmation of intrahepatic cholangiocarcinoma (iCCA)
* The following tumor characteristics must be met

  * Unresectable disease: HCC (group 2) or intrahepatic CCA (group 3)
  * Measurable or evaluable disease
  * All lesions should be treatable by EBRT while meeting normal tissue constraints
  * Tumor lesions should be accessible using an ultrasound (US)-guided approach for intratumoral DC injection
  * No evidence of extrahepatic tumor (excluding tumor thrombus) by computed tomography (CT) or magnetic resonance imaging (MRI) scan

    * NOTE: Patients who are not candidates for surgical treatment or for ablation with curative intent are allowed
* Good candidate for standard of care high-dose conformal EBRT in the view of the investigator
* Eastern Cooperative Oncology Group (ECOG) performance status (PS) 0 or 1
* GROUP 2 HCC ONLY: Absolute neutrophil count (ANC) >= 1000/mm^3 (obtained =< 15 days prior to registration)
* GROUP 2 HCC ONLY: Absolute lymphocyte count (ALC) >= 500/mm^3 (obtained =< 15 days prior to registration)
* GROUP 2 HCC ONLY: Absolute monocyte count (AMC) >= 300/mm^3 (obtained =< 15 days prior to registration)
* GROUP 2 HCC ONLY: Platelet count >= 50,000/mm^3 (obtained =< 15 days prior to registration)
* GROUP 2 HCC ONLY: Hemoglobin >= 9.0 g/dL (obtained =< 15 days prior to registration)
* GROUP 2 HCC ONLY: Total bilirubin < 1.5 mg/dL (obtained =< 15 days prior to registration)
* GROUP 2 HCC ONLY: Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) =< 5 x upper limit of normal (ULN) (obtained =< 15 days prior to registration)
* GROUP 2 HCC ONLY: Creatinine =< 2 mg/dL (obtained =< 15 days prior to registration)
* GROUP 2 HCC ONLY: Prothrombin time (PT)/international normalized ratio (INR)/activated partial thromboplastin time (aPTT) =< 1.5 x ULN (obtained =< 15 days prior to registration)
* GROUP 2 HCC ONLY: Absence of proteinuria at screening as demonstrated by one of the following:

  * Urine protein/creatinine (UPC) ratio < 1.0 at screening OR
  * Urine dipstick for proteinuria < 2+ (patients discovered to have >= 2+ proteinuria on dipstick urinalysis at baseline should undergo a 24-hour urine collection and must demonstrate =<1g of protein in 24 hours to be eligible)
* GROUP 3 iCCA ONLY: Absolute neutrophil count (ANC) ≥ 1500/mm^3 (obtained =< 15 days prior to registration)
* GROUP 3 iCCA ONLY: Absolute lymphocyte count ≥ 500/mm^3 (obtained =< 15 days prior to registration)
* GROUP 3 iCCA ONLY: Absolute monocyte count ≥ 300/mm^3 (obtained =< 15 days prior to registration)
* GROUP 3 iCCA ONLY: Platelet count ≥ 100,000/mm^3 (obtained =< 15 days prior to registration)
* GROUP 3 iCCA ONLY: Hemoglobin ≥ 9.0 g/dL (obtained =< 15 days prior to registration)
* GROUP 3 iCCA ONLY: Total bilirubin < 1.5 x ULN (obtained =< 15 days prior to registration)
* GROUP 3 iCCA ONLY: Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) and alkaline phosphatase (ALP) ≤ 2.5 x ULN (obtained =< 15 days prior to registration)
* GROUP 3 iCCA ONLY: Creatinine ≤ 2 mg/dL (obtained =< 15 days prior to registration)
* GROUP 3 iCCA ONLY: Serum albumin ≥ 25 g/L (2.5 g/dL) (obtained =< 15 days prior to registration)
* GROUP 3 iCCA ONLY: PT/INR/aPTT ≤ 1.5 x ULN (obtained =< 15 days prior to registration)

  * NOTE: If patient is receiving therapeutic anticoagulation, patient must be on a stable anticoagulant regimen
* GROUP 3 iCCA ONLY: Calcium ≤ 12 mg/dl or corrected serum calcium ≤ ULN (obtained =< 15 days prior to registration)
* Negative pregnancy test done =< 8 days prior to registration, for persons of childbearing potential only
* GROUP 3 ONLY: Negative hepatitis B surface antigen (HBsAg) test at screening
* GROUP 3 ONLY: Negative hepatitis C virus antibody (HCV Ab) test at screening, or positive HCV antibody test followed by a negative HCV ribonucleic acid (RNA) test at screening. (NOTE: HCV RNA test will be performed only for patients who have a positive HCV antibody test.)
* Ability to provide written consent
* Willingness to return to enrolling institution for follow-up (during the active monitoring phase of the study)
* Willingness to provide blood and tissue samples for correlative research purposes

Exclusion Criteria:

* Any of the following because this study involves an investigational agent, the genotoxic, mutagenic and teratogenic effects of which on the developing fetus and newborn are unknown:

  * Pregnant persons
  * Nursing persons
  * Persons of childbearing potential who are unwilling to employ highly effective contraception during heterosexual intercourse while on this study and for 5 months after the last dose of study medication
* Co-morbid systemic illnesses or other severe concurrent disease which, in the judgment of the investigator, would make the patient inappropriate for entry into this study or interfere significantly with the proper assessment of safety and toxicity of the prescribed regimens
* Immunocompromised patients and patients known to be HIV positive.

  * NOTE: Patients known to be HIV positive, but without clinical evidence of an immunocompromised state, are eligible for this trial if they are stable on anti-retroviral therapy, have a CD4+ T cell count ≥ 200/uL, and have an undetectable viral load
* Uncontrolled intercurrent illness including, but not limited to:

  * Ongoing or active infection requiring systemic treatment or that could impact patient safety
  * Severe infection ≤ 4 weeks prior to registration, including, but not limited to, hospitalization for complications of infection, bacteremia, or severe pneumonia
  * Significant cardiovascular disease (New York Heart Association [NYHA] class II), symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia
  * Or, psychiatric illness/social situations (e.g., substance abuse) that would limit compliance with study requirements
* Receiving any other investigational agent that would be considered a treatment for the primary neoplasm
* Other active malignancy =< 1 year prior to registration that is considered by the investigator to interfere with the current treatment or measurement of outcomes
* Major surgery =< 4 weeks prior to enrollment (other than diagnostic surgery or surgical spacer placement in preparation for radiation treatment), or anticipation of need for a major surgical procedure during the study
* History of hypersensitivity or anaphylactoid reactions to pneumococcal vaccine or any component of the formulation, including diphtheria toxoid
* Active or history of autoimmune disease or immune deficiency, including but not limited to,myasthenia gravis, myositis, autoimmune hepatitis, Crohn's disease, inflammatory bowel disease, antiphospholipid antibody syndrome, rheumatoid arthritis, Sjogren syndrome, systemic lupus erythematosus, Guillain-Barre syndrome, multiple sclerosis, Wegener granulomatosis, or similar conditions

  * NOTE: Exceptions are allowed for:

    * Patients with hypothyroidism on thyroid replacement therapy
    * Patients with type 1 diabetes mellitus on insulin regimen
    * Patients with eczema, psoriasis lichen simplex chronicus, or vitiligo with dermatologic manifestations only (e.g., patients with psoriatic arthritis are excluded) are eligible for the study provided all of the following conditions are met:

      * Rash must cover < 10% of body surface area
      * Disease is well controlled at baseline and requires only low-potency topical corticosteroids
      * There has been no occurrence of acute exacerbations of the underlying condition requiring psoralen plus ultraviolet A radiation, methotrexate, retinoids, biologic agents, oral calcineurin inhibitors, or high potency or oral corticosteroids ≤ 12 months prior to registration
* Requires anticoagulant treatment (INR > 1.5 x ULN) or use of anti-platelet agents that cannot be discontinued for the intratumoral injection procedure

  * NOTE: Heparin for line patency without detectable lab abnormalities in coagulation will be allowed
* Corticosteroids =< 2 weeks prior to registration, including oral, intravenous (IV), subcutaneous, or inhaled routes of administration

  * NOTE: Patients on chronic corticosteroids for adrenal insufficiency or other reasons may enroll if they receive less than 10 mg/day of prednisone (or equivalent)
  * NOTE: Exception allowed for patients who need prophylactic steroids prior to imaging for contrast allergies

    * Exception: Patients who received acute, low-dose systemic immunosuppressant medication or a one-time pulse dose of systemic immunosuppressant medication (e.g., 48 hours of corticosteroids for a contrast allergy) are eligible for the study
    * Exception: Patients who received mineralocorticoids (e.g., fludrocortisone), corticosteroids for chronic obstructive pulmonary disease (COPD) or asthma, or low-dose corticosteroids for orthostatic hypotension or adrenal insufficiency are eligible for the study
* History of myocardial infarction =< 6 months, or congestive heart failure requiring use of ongoing maintenance therapy for life-threatening ventricular arrhythmias
* Child Pugh class B or C cirrhosis of the liver
* Previously received immune modulating therapies including but not limited to immune checkpoint inhibitors targeting PD-1 PDL-1 CTLA4, etc.; or prior dendritic cell therapy
* Prior liver radiation, including radioembolization
* GROUP 2 ONLY: Barcelona Clinic Liver Cancer (BCLC) stage D disease
* GROUP 2 ONLY: History of untreated high-risk gastroesophageal varices
* GROUP 3 ONLY: History of idiopathic pulmonary fibrosis, organizing pneumonia (e.g., bronchiolitis obliterans), drug-induced pneumonitis, or idiopathic pneumonitis, or evidence of active pneumonitis
* Active tuberculosis
* Treatment with therapeutic oral or IV antibiotics ≤ 2 weeks prior to registration

  * NOTE: Exception for patients receiving prophylactic antibiotics (e.g., to prevent a urinary tract infection or chronic obstructive pulmonary disease exacerbation) are eligible for the study
* Prior allogeneic stem cell or solid organ transplantation
* Treatment with a live, attenuated vaccine ≤ 4 weeks prior to registration, or anticipation of need for such a vaccine during study treatment, within 90 days after the final dose of tiragolumab, or within 5 months after the final dose of atezolizumab

  * NOTE: Patients being treated with chemotherapy (e.g., carboplatin, cisplatin, pemetrexed, paclitaxel, or gemcitabine) should not receive live vaccines
* GROUP 3 ONLY: Acute Epstein-Barr virus (EBV) infection or known or suspected chronic active EBV at screening

  * NOTE: Patients with symptoms such as splenomegaly, fever, sore throat, non-malignant cervical lymphadenopathy, and/or tonsillar exudate, should undergo an EBV polymerase chain reaction (PCR) test to screen for acute infection or suspected chronic active infection. Patients with a positive EBV PCR test are excluded. Patients with positive Epstein-Barr virus (EBV) viral capsid antigen immunoglobulin M (IgM) test at screening are excluded
* GROUP 3 ONLY: History of severe allergic anaphylactic reactions to chimeric or humanized antibodies or fusion proteins
* GROUP 3 ONLY: Known hypersensitivity to Chinese hamster ovary cell products or to any component of the atezolizumab or tiragolumab formulation
* GROUP 3 ONLY: Known allergy or hypersensitivity to any component of the chemotherapy regimen the patient may receive during the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 85 (Estimated)
Dates: Start 2019-09-19 (Actual); Primary Completion 2027-08-31 (Estimated); Study Completion 2028-02-29 (Estimated)

PRIMARY OUTCOMES:
Incidence of significant toxicity (Pilot study) | Up to completion of cycle 2 (each cycle is 28 days)
  A significant toxicity is defined as a dose limiting toxicity that is possibly, probably, or definitely related to dendritic cell (DC) treatment. Toxicities will be assessed using the Cancer Therapy Evaluation Program active version of the Common Terminology Criteria for Adverse Events.
Progression-free survival rate at 2 years (Phase II) | At 2 years
  Defined as the time from registration to disease progression or death due to all causes.
PFS (Phase II Group 3) | Up to 5 years
  Defined as the time from registration to disease progression or death due to all causes.

SECONDARY OUTCOMES:
Overall response rate | Up to 1 year post treatment
  The overall response rate will be estimated by the number of patients with an objective status of complete response (CR) or partial response (PR) divided by the total number of evaluable patients. Exact binomial 95% confidence intervals for the true overall response rate will be calculated.
Number of patients who received at least one dose of intratumoral DC injection | Up to 1 year post treatment
  The feasibility of the regimen will be estimated by the number of patients who received at least one dose of intratumoral DC injection divided by the total number of patients who received apheresis.
Clinical benefit rate | Up to 1 year post treatment
  The clinical benefit rate will be estimated by the number of patients with an objective status of stable disease or CR or PR at any time divided by the total number of evaluable patients. Exact binomial 95% confidence intervals for the true clinical benefit rate will be calculate
Time to response | Up to 1 year post treatment
  Time to response is defined for all evaluable patients who have achieved an objective response as the date of initiation of vaccination treatment to the date at which the patient's objective status is first noted to be either a CR or PR. Time to response will be summarized descriptively using Kaplan-Meier methodology.
Duration of response | Up to 1 year post treatment
  Duration of response is defined for all evaluable patients who have achieved an objective response as the date at which the patient's objective status is first noted to be either a CR or PR to the earliest date progression is documented. Duration of response will be summarized descriptively using Kaplan-Meier methodology.
Overall survival | Up to 5 years
  Defined as the time from registration to death from any cause.
Progression-free survival | Up to 5 years
  Defined as the time from registration to disease progression or death due to all causes.

OTHER OUTCOMES:
Change in target lesion measurements | Baseline up to 1 year post treatment
  All enhancing lesions will be evaluated over time for each patient. The percent change from baseline in target lesion measurements will be assessed over time. Differences in values over time will be summarized descriptively and graphically.
Change in immunologic correlates before and after vaccination treatment | Baseline up to 1 year post treatment
  Change in immunologic correlates before and after vaccination treatment will be evaluated and summarized both quantitatively and graphically. Each of the correlative endpoints will be summarized individually, but will also be evaluated in terms of their relationships to one another; i.e., will use Spearman rank correlation coefficient to assess the correlations between baseline levels as well as between changes before and after treatment in these immunologic markers. In addition, these immunologic markers will be correlated with cancer and treatment related outcomes (e.g. response, adverse events). Relationships will also be explored graphically using scatter plots.

CONTACTS AND LOCATIONS:
Overall Officials: Lewis R. Roberts, MD, PhD, Principal Investigator — Mayo Clinic in Rochester
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials